CLINICAL TRIAL: NCT05553600
Title: An Open-Label Clinical Validation Study of an Applicator Tampon
Brief Title: Tampon Design Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AFC-21-001
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Menstruation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Regular Absorbency (Other): Modified regular absorbency tampon versus regular absorbency reference tampon
  Interventions: Device: Tampon BR; Device: Tampon CR
- Super Absorbency (Other): Modified super absorbency tampon versus super absorbency reference tampon
  Interventions: Device: Tampon BS; Device: Tampon CS

INTERVENTIONS:
Device: Tampon BR — Modified Regular Absorbency Tampons
  Arms: Regular Absorbency
Device: Tampon CR — Reference Regular Absorbency Tampons
  Arms: Regular Absorbency
Device: Tampon BS — Modified Super Absorbency Tampons
  Arms: Super Absorbency
Device: Tampon CS — Reference Super Absorbency Tampons
  Arms: Super Absorbency

SUMMARY:
This prospective multi-center, open-label, randomized, cross-over study is designed to validate the user needs of a tampon design. The hypothesis is that user needs are met.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to read and provide written informed consent.
* Female in good general health, age 18-49 (inclusive).
* History of regular menstrual cycles during the previous 3months lasting approximately 21-35 days, including at least 4 days of menstruation, and expecting to menstruate during the study period.
* History of use of applicator tampons without discomfort.
* Normally use at least 6 tampons for protection during menstruation.
* Normally uses regular, super, and/or super plus absorbency tampons for menstrual protection.
* Agrees to the conduct of all study procedures, including gynecological exams (if applicable), and agrees to follow all study instructions and return for scheduled appointments.
* Has used an acceptable form of birth control for at least one month prior to enrollment and for the duration of the study.

Key Exclusion Criteria:

* Pregnant, lactating or is trying to become pregnant.
* Less than six (6) weeks post-partum.
* Has a menstrual abnormality (such as oligomenorrhea or amenorrhea).
* Has a known allergy or sensitivity to components of the investigational products, including rayon.
* Any other medical condition or history, as determined by the Investigator that could compromise the study results or subject safety.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 732 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Velocity Clinical Research, Boise, Idaho
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - Princeton Consumer Research, Raritan, New Jersey
  - Velocity Clinical Research, Anderson, South Carolina
  - Velocity Clinical Research, Greenville, South Carolina
  - Signature Gyn Services, Fort Worth, Texas
  - TMC Life Research, Inc., Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 732 subjects enrolled were assigned to a study arm.
Groups:
- Regular Absorbency: BR, Then CR: Participants received tampon code BR (modified regular absorbency tampon) to use during their first menstrual cycle, followed by tampon code CR (regular absorbency reference tampon) to use for their second menstrual cycle.
- Regular Absorbency: CR, Then BR: Participants received tampon code CR (regular absorbency reference tampon) to use during their first menstrual cycle, followed by tampon code BR (modified regular absorbency tampon) to use for their second menstrual cycle.
- Super Absorbency: BS, Then CS: Participants received tampon code BS (modified super absorbency tampon) to use during their first menstrual cycle, followed by tampon code CS (super absorbency reference tampon) to use for their second menstrual cycle.
- Super Absorbency: CS, Then BS: Participants received tampon code CS (super absorbency reference tampon) to use during their first menstrual cycle, followed by tampon code BS (modified super absorbency tampon) to use for their second menstrual cycle.
Period: Prior to First Menstrual Cycle Starting
Arm/Group | Regular Absorbency: BR, Then CR | Regular Absorbency: CR, Then BR | Super Absorbency: BS, Then CS | Super Absorbency: CS, Then BS
Started | 201 | 203 | 166 | 162
Completed | 174 | 173 | 145 | 140
Not Completed | 27 | 30 | 21 | 22
Not completed — Withdrawal by Subject | 4 | 8 | 6 | 7
Not completed — Protocol Violation | 0 | 1 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 16 | 13 | 12 | 10
Not completed — Other various reasons | 7 | 8 | 3 | 2
Period: Prior to Second Menstrual Cycle Starting
Arm/Group | Regular Absorbency: BR, Then CR | Regular Absorbency: CR, Then BR | Super Absorbency: BS, Then CS | Super Absorbency: CS, Then BS
Started | 174 | 173 | 145 | 140
Completed | 156 | 151 | 132 | 121
Not Completed | 18 | 22 | 13 | 19
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 1
Not completed — Protocol Violation | 1 | 3 | 0 | 1
Not completed — Physician Decision | 6 | 4 | 1 | 6
Not completed — Lost to Follow-up | 5 | 6 | 4 | 3
Not completed — Other various reasons | 4 | 7 | 3 | 8
Period: After Second Menstrual Cycle Began
Arm/Group | Regular Absorbency: BR, Then CR | Regular Absorbency: CR, Then BR | Super Absorbency: BS, Then CS | Super Absorbency: CS, Then BS
Started | 156 | 151 | 132 | 121
Completed | 155 | 151 | 132 | 121
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular Absorbency | Super Absorbency | Total
Number analyzed (Participants) | 404 | 328 | 732
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (8.11) | 34.6 (7.62) | 33.6 (7.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 404 | 328 | 732
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 56 | 137
  Not Hispanic or Latino | 318 | 264 | 582
  Unknown or Not Reported | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 17 | 10 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 115 | 123 | 238
  White | 264 | 185 | 449
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Used Tampons That Have Elongated
Description: The percentage of used tampons within each test code that have elongated >10mm. The denominator for the percentage calculation is based upon the number of used tampons returned within each test code.
Time Frame: At the end of 1 menstrual period (up to 10 days) for each intervention
Population: All subjects who have no major protocol deviations and return at least 1 tampon that can be assessed for elongation.
Measure: Count of Units; unit: tampons
Units Other Than Participants: tampons
Groups:
- Tampon BR: Modified regular absorbency tampon
- Tampon CR: Reference regular absorbency tampon
- Tampon BS: Modified super absorbency tampon
- Tampon CS: Reference super absorbency tampon
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
Number analyzed (Participants) | 264 | 264 | 223 | 222
Number analyzed (tampons) | 2635 | 2577 | 2454 | 2410
tampons | 2 | 75 | 4 | 48

2. Secondary Outcome: Validation of Performance User Needs Based on Participant Diary Responses.
Description: Percentage of participants reporting tampons performed as needed through diary responses. The following responses were solicited once at the end of the menstrual period.
Time Frame: At the end of 1 menstrual period (up to 10 days) for each intervention
Population: All subjects randomized into the study
Measure: Count of Participants; unit: Participants
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
Number analyzed (Participants) | 322 | 321 | 260 | 266
Participants
  Participants reporting they were able to open the box and retrieve the wrapped tampons | 322 | 320 | 260 | 266
  Participants reporting they were able to open each tampon wrapper | 321 | 319 | 260 | 266
  Participants reporting tampons were clean prior to use | 322 | 320 | 260 | 266
  Participants reporting they were able to insert the tampons with applicator | 297 | 295 | 238 | 249

3. Secondary Outcome: Validation of Performance User Needs Based on Participant Diary Responses
Description: Percentage of tampons performing as needed. The following diary responses were solicited after every tampon use.
Time Frame: At the end of 1 menstrual period (up to 10 days) for each intervention
Population: All subjects randomized into the study
Measure: Count of Units; unit: Tampons
Units Other Than Participants: Tampons
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
Number analyzed (Participants) | 323 | 323 | 263 | 268
Number analyzed (Tampons) | 3234 | 3141 | 2907 | 2877
Tampons
  Tampons that remained white when subject was experiencing flow: number analyzed (Tampons) | 3187 | 3086 | 2871 | 2831
  Tampons that remained white when subject was experiencing flow | 38 | 33 | 43 | 20
  Tampons participants reported they were able to remove | 3227 | 3133 | 2904 | 2870

4. Secondary Outcome: Validation of Packaging/Labeling User Needs Based on Interview Responses
Description: Proportion of participants able to locate key packaging/labeling information.
Time Frame: At baseline, prior to any interventions
Population: All subjects randomized into the study and the gynecological exam subset. Packaging interview was conducted at the baseline visit, independent of and prior to any intervention. Therefore, results are broken out by study arm. Responses for some questions were not recorded for all subjects due to protocol deviations.
Measure: Count of Participants; unit: Participants
Groups:
- Packaging Interview Group: Subset of the total population that agreed to participate in pre- and post-use gynecological exams and a packaging and labeling interview
Arm/Group | Packaging Interview Group
Number analyzed (Participants) | 147
Participants
  Able to identify tampon absorbency on regular absorbency box | 146
  Able to identify tampon absorbency on super absorbency box | 146
  Able to identify tampon absorbency on super plus absorbency box | 146
  Able to identify tampon absorbencies on multipack box: number analyzed (Participants) | 140
  Able to identify tampon absorbencies on multipack box | 139
  Able to identify tampon absorbency ranges for entire line on box | 147
  Able to identify toxic shock syndrome warning on box | 147
  Able to identify how long a tampon should be used on box | 132
  Able to identify regular absorbency wrapped tampon: number analyzed (Participants) | 140
  Able to identify regular absorbency wrapped tampon | 138
  Able to identify super absorbency wrapped tampon: number analyzed (Participants) | 140
  Able to identify super absorbency wrapped tampon | 140
  Able to identify super plus absorbency wrapped tampon: number analyzed (Participants) | 140
  Able to identify super plus absorbency wrapped tampon | 139
  Able to identify instructions for use on insert: number analyzed (Participants) | 146
  Able to identify instructions for use on insert | 146
  Able to identify toxic shock syndrome information on insert: number analyzed (Participants) | 146
  Able to identify toxic shock syndrome information on insert | 144

5. Secondary Outcome: Number of Subjects That Had Any Lesions Noted During Gynecological Exam
Description: Number of subjects noted during pre- and post-use gynecological exams that had any lesions by anatomical location
Time Frame: Within 72 hours prior expected menstruation (pre-use) and within 72 hours after last tampon use (post-use) for each intervention
Population: All subjects randomized into the study and participating in the gynecological exam subset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
Number analyzed (Participants) | 68 | 63 | 50 | 54
Participants
  Perineum : Pre-Use | 0 | 1 | 0 | 0
  Perineum : Post-Use | 1 | 0 | 0 | 0
  Vulva : Pre-Use | 0 | 1 | 1 | 1
  Vulva : Post-Use | 0 | 0 | 0 | 2
  Urethra : Pre-Use | 0 | 0 | 0 | 0
  Urethra : Post-Use | 0 | 0 | 0 | 0
  Vagina : Pre-Use | 0 | 0 | 0 | 0
  Vagina : Post-Use | 0 | 0 | 0 | 0
  Cervix : Pre-Use | 0 | 0 | 0 | 0
  Cervix : Post-Use | 0 | 1 | 0 | 0

6. Secondary Outcome: Additional Gynecological Exam Results: Pre-use Vaginal pH
Description: Vaginal pH prior to tampon use.
Time Frame: as for outcome 5
Population: All subjects randomized into the study and participating in the gynecological exam subset that had pre-use pH readings.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
Number analyzed (Participants) | 62 | 62 | 48 | 53
pH | 4.81 (0.436) | 4.72 (0.380) | 4.99 (0.672) | 5.14 (0.805)

7. Secondary Outcome: Additional Gynecological Exam Results: Post-use Vaginal pH
Description: Vaginal pH after tampon use.
Time Frame: as for outcome 5
Population: All subjects randomized into the study and participating in the gynecological exam subset that had post-use pH readings.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
Number analyzed (Participants) | 65 | 57 | 48 | 54
pH | 4.85 (0.499) | 4.76 (0.412) | 5.19 (0.848) | 4.86 (0.518)

8. Secondary Outcome: Additional Gynecological Exam Results: Number of Participants With Suspected Infections, Other Abnormal Findings, and Clinically Significant Results
Description: Additional gynecological exam results prior to and following tampon use including: number of participants with suspected infections, other abnormal finding, and exam results that the investigators found clinically significant.
Time Frame: as for outcome 5
Population: All subjects randomized into the study and participating in the gynecological exam subset.
Measure: Count of Participants; unit: Participants
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
Number analyzed (Participants) | 68 | 63 | 50 | 54
Participants
  Suspected Infection : Pre-Use | 0 | 0 | 1 | 0
  Suspected Infection : Post-Use | 6 | 0 | 2 | 1
  Other abnormal finding : Pre-Use | 0 | 1 | 0 | 0
  Other abnormal finding : Post-Use | 1 | 0 | 0 | 0
  Clinically significant exam results : Pre-Use | 0 | 0 | 0 | 0
  Clinically significant exam results : Post-Use | 5 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 months
Arm/Group | Tampon BR | Tampon CR | Tampon BS | Tampon CS
All-Cause Mortality (participants affected / at risk) | 0/323 | 0/323 | 0/263 | 0/268
Serious Adverse Events (participants affected / at risk) | 1/323 | 0/323 | 0/263 | 0/268
Other Adverse Events (participants affected / at risk) | 0/323 | 0/323 | 0/263 | 0/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tampon BR (N=323) | Tampon CR (N=323) | Tampon BS (N=263) | Tampon CS (N=268)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT05553600/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT05553600/SAP_001.pdf